CLINICAL TRIAL: NCT07023458
Title: The Effects of Hypoxic Burden on Executive Function (EF) in Preschool Children With Obstructive Sleep Apnea
Status: Not yet recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sarisa Thawongit, Principal Investigator, Mahidol University
Other Study IDs: COA119/2025
Record Dates: First submitted 2025-06-07; First posted 2025-06-17 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: All participants in the group will undergo polysomnography, Denver test and BRIEF-P test for executive function
  Interventions: Diagnostic Test: Brief-P

INTERVENTIONS:
Diagnostic Test: Brief-P — Executive function test in preschool children with OSA

SUMMARY:
The goal of this observational study is to study the effect of hypoxic burden on executive function in preschool children aged 2-6 years who have OSA.

The main question it aims to answer is Effect of hypoxic burden from OSA to executive function measured by BRIEF-P in preschool children..

DETAILED DESCRIPTION:
There is no comparison group in this study Participants will performed full night polysomnography, Denver and BRIEF-P test within 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-6 years old with OSA

Exclusion Criteria:

* Underlying diseases : hypoventilation, neuromuscular diseases, etc.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Siriraj Hospital
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Executive function from BRIEF-P test | 3 months
  T-scores at or below 59 are considered to be within the typical range

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand